CLINICAL TRIAL: NCT01214655
Title: Phase 1 Study of LY2523355 in Patients With Acute Leukemia
Brief Title: A Study for Patients With Acute Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Primary objective has been met in the absence of clinically meaningful remissions
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12119; I1Y-MC-JFBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-01; First posted 2010-10-05 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2017-09

CONDITIONS: Acute Leukemia
Keywords: Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia,Blast Crisis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis | interventions — litronesib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2523355 on Days 1, 2, and 3 (Experimental): Starting dose was 2 milligrams per meter squared (mg/m^2) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day Cycle.
  Interventions: Drug: LY2523355
- LY2523355 on Days 1, 5, and 9 (Experimental): Starting dose was 8 milligrams per meter squared (mg/m^2) administered by a 1-hour IV infusion over 1 hour on Days 1, 5, and 9 of every 21-day Cycle.
  Interventions: Drug: LY2523355

INTERVENTIONS:
Drug: LY2523355 — Administered as a 1-hour IV infusion for at least 2 cycles. Cycle length is 21 days. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion is met.

SUMMARY:
This study is a multicenter, nonrandomized, open-label, dose-escalation with intra-patient dose-escalation, Phase 1 study of intravenous LY2523355 to determine the dose of LY2523355 that can be safely administered to participants with acute leukemia. Part A and Part B are dose escalation of two schedules in participants with acute leukemia. Parts A and B will enroll concurrently. Part C is a dose expansion for each schedule in participants with acute myeloblastic leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

Dose escalation period for both schedules:

* Participants must have a confirmed diagnosis of acute leukemia regardless of sub-type and for whom experimental Phase 1 therapy is appropriate.
* Are greater than or equal to 18 years of age.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Females with childbearing potential must have had a negative urine or serum pregnancy test less than or equal to 7 days prior to the first dose of study drug.

Dose confirmation period for both schedules:

* Participant must have a confirmed diagnosis of untreated acute myeloblastic leukemia (AML), should not be a candidate for standard therapy, and a clinical trial is a preferred treatment option or have acute AML that is relapsed or refractory to no more than 2 prior induction regimens. Hydroxyurea to control prior blast counts is not considered a prior regimen.
* Are greater than or equal to 60 years of age.
* Have a performance status of 0 or 1 on the ECOG scale.
* Females with childbearing potential must have had a negative urine or serum pregnancy test less than or equal to 7 days prior to the first dose of study drug.

Exclusion Criteria:

* Have received treatment within 28 days of the initial dose of study drug with a drug that has not received regulatory approval for any indication.
* Participants with known central nervous system (CNS) leukemia by spinal fluid cytology or imaging. A lumbar puncture is not required unless CNS involvement is clinically suspected. Participants with signs or symptoms of leukemic meningitis or a history of leukemic meningitis must have a negative lumbar puncture within 2 weeks of study enrollment.
* Have other active malignancy (with the exception of basal and squamous cell skin cancer) at time of study entry.
* Have had an autologous or allogenic bone marrow transplant within 3 months. All organ toxicity must be resolved.
* Have evidence of graft-versus-host disease due to an allogenic bone marrow transplant.
* Have uncontrolled systemic infection.
* Females who are pregnant or lactating.
* Have known positive test results in human immunodeficiency virus (HIV), hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb) (screening not required).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A participant was considered to have completed the trial if they received at 2 cycles of treatment. Participant Flow Arms represent schedule of dosing, with dose escalation, dose levels and participants who joined the dose level presented as Milestones. Study was based on best Schedule of dosing, not dose levels.
Groups:
- Schedule A LY2523355: Participants received a dose escalation to maximum tolerated dose (MTD) from 2 mg/m²/day to 4,5 and 6 mg/m²/day during a 1 hour (hr) infusion on Days 1,2, 3 (Schedule A) of a 21 day cycle. Participants did not have to escalate doses and participants could join at a higher dose level.
- Schedule B LY2523355: Participants received a dose escalation to maximum tolerated dose (MTD) ranging from 8 mg/m²/day (starting dose) to 10,12 and 14 mg/m²/day during a 1 hour (hr) infusion on Days 1,5, 9 (Schedule B)of a 21 day cycle Participants did not have to escalate doses and participants could join at a higher dose level.
- Schedule C LY2523355: Starting dose was 5 mg/m²/day administered by IV infusion over 1 hour on Days 1, 2, and 3 (Schedule C) of every 21-day Cycle.
Period: Part A
Arm/Group | Schedule A LY2523355 | Schedule B LY2523355 | Schedule C LY2523355
Started | 10 (Total on Schedule A, dose days 1,2,3) | 0 | 0
Received 2 mg Study Drug | 3 | 0 | 0
Escalated From 2 to 4 mg/m²/Day | 3 | 0 | 0
Joined 4 mg Group (4 participants received 4 mg/m²/day) | 1 | 0 | 0
Escalated From 4 mg Study Drug | 0 | 0 | 0
Joined 5 mg Study Drug (2 participants received 5 mg/m²/day) | 2 | 0 | 0
Escalated From 5 mg Study Drug | 1 | 0 | 0
Joined 6 mg Group | 4 | 0 | 0
Received 6 mg Study Drug | 5 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 8 | 0 | 0
Not completed — Progressive Disease | 7 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Part B
Arm/Group | Schedule A LY2523355 | Schedule B LY2523355 | Schedule C LY2523355
Started | 0 (Part A participants did not enroll in Part B. Participants in A, B, C are considered Cohorts.) | 15 (Total on Schedule B, dose days 1,5,9) | 0
Received at Least 1 Dose of Study Drug | 0 | 15 | 0
Recieved 8 mg/m²/Day Study Drug | 0 | 4 | 0
Escalated From 8 to 10 mg/m²/Day | 0 | 2 | 0
Joined 10 mg/m²/Day Study D (5 participants received 10 mg/m²/day Study Drug) | 0 | 3 | 0
Escalated to 12 mg/m²/Day | 0 | 2 | 0
Joined 12 mg/m²/Day (7 participants received 12 mg/m²/day Study Drug) | 0 | 5 | 0
Escalated From 12 to 14 mg/m²/Day | 0 | 1 | 0
Joined 14 mg/m²/Day (4 participants received 14 mg/m²/day Study Drug) | 0 | 3 | 0
Completed | 0 | 2 | 0
Not Completed | 0 | 13 | 0
Not completed — Progressive disease | 0 | 10 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Period: Part C
Arm/Group | Schedule A LY2523355 | Schedule B LY2523355 | Schedule C LY2523355
Started | 0 | 0 | 8 (Total on Schedule C, dose days 1,2,3)
Received at Least 1 Dose of 5 mg/m²/Day | 0 | 0 | 8
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 7
Not completed — Progressive Disease | 0 | 0 | 5
Not completed — Death | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study medication (LY2523355).
Groups:
- Schedule A LY2523355: Starting dose was 2 milligrams per meter squared per day (mg/m^2/day) administered by intravenous (IV) infusion over 1 hour on Days 1, 2, and 3 of every 21-day Cycle.
- Schedule B LY2523355: Starting dose was 8 mg/m^2/day administered by IV infusion over 1 hour on Days 1, 5, and 9 of every 21-day Cycle.
- Schedule C LY2523355: Starting dose was 5 mg/m^2/day administered by IV infusion over 1 hour on Days 1, 2, and 3 of every 21-day Cycle.
  No participants in Part C escalated from their initial dose.
- Total: Total of all reporting groups
Arm/Group | Schedule A LY2523355 | Schedule B LY2523355 | Schedule C LY2523355 | Total
Number analyzed (Participants) | 10 | 15 | 8 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (19.43) | 65.3 (12.98) | 70.7 (5.75) | 66.0 (13.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 5 | 14
  Male | 4 | 12 | 3 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 7 | 14 | 7 | 28
  African | 2 | 0 | 1 | 3
  Hispanic | 0 | 1 | 0 | 1
  Native American | 0 | 0 | 0 | 0
  East Asian | 1 | 0 | 0 | 1
  West Asian | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 15 | 8 | 33
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death) as follows: 0 - Fully Active; 1 - Ambulatory, Restricted Strenuous Activity; 2 - Ambulatory, No Work Activities; 3 - Partially Confined to Bed, Limited Self Care; 4 - Completely Disabled; and 5 - Dead.
  Participants
    ECOG Status 0 | 6 | 2 | 1 | 9
    ECOG Status 1 | 4 | 7 | 6 | 17
    ECOG Status 2 | 0 | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose and Schedule for Phase 2 Studies in Acute Leukemia
Description: The recommended dose and schedule for Phase 2 studies of LY2523355 with acute leukemia was determined by a modification of the continual reassessment method. The sample size to adequately determine the maximum tolerated dose (MTD) for both schedules in this study was a function of a priori estimates for the dose-toxicity relationship as well as the initial dose in each schedule, the rate of dose escalation, and the observed dose-toxicity relationship. Before MTD could be determined for Part B (Days 1, 5, and 9 of a 21-day cycle), this study was paused for futility analysis.
Time Frame: Baseline up to the end of Cycle 2 (Day 42)
Population: Participants who received at least one dose of study medication (LY2523355).
Measure: Number; unit: mg/m^2/day; Days 1, 2, and 3
Groups:
- LY2523355: Escalating doses starting at 2 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day Cycle in Part A of the study. Escalating doses starting at 8 mg/m^2/day administered by a 1-hour IV infusion on Days 1, 5, and 9 of every 21-day Cycle in Part B of the study. Dose of 5 mg/m^2/day administered by a 1-hour IV infusion on Days 1, 2, and 3 of every 21-day Cycle in Part C of the study.
Arm/Group | LY2523355
Number analyzed (Participants) | 33
mg/m^2/day; Days 1, 2, and 3 | 5

2. Secondary Outcome: Number of Participants With Clinically Significant Effects
Description: Clinically significant effects were defined as serious and other non-serious adverse events (AEs).
  A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline up to study completion (up to 213 days)
Population: Participants who received at least one dose of study medication (LY2523355).
Measure: Count of Participants; unit: Participants
Groups:
- Schedule A LY2523355: Escalating doses starting at 2 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day Cycle in Part A of the study.
- Schedule C LY2523355: Starting dose was 5 mg/m^2/day administered by IV infusion over 1 hour on Days 1, 2, and 3 of every 21-day Cycle.
Arm/Group | Schedule A LY2523355 | Schedule B LY2523355 | Schedule C LY2523355
Number analyzed (Participants) | 10 | 15 | 8
Participants | 7 | 9 | 4

3. Secondary Outcome: Pharmacokinetics, Maximum Plasma Concentration (Cmax), Single Dose
Description: The maximum plasma concentration (Cmax) was the maximum plasma concentration obtained from the plasma concentration versus time curves of LY2523355 were calculated to assess intra and intercycle variability, depending on dosage cycle.
Time Frame: Cycle 1(Day 1),: Predose, 1 hour (hr), 2 hr, 3 hr, 4 hr, 6 hr, 8, hr, 12 hr, 24 hr, 48 hr, 72 hr postdose
Population: Participants who received one dose of LY2523355 on Day 1 of Cycle 1(Schedule A,B,C) with evaluable pharmacokinetic data to enable determination of the LY2523355 plasma Cmax on Day 1. Schedule A,C data was combined for 5 mg, 2 participants received and incorrect dose of 6 mg and 16 mg are included in data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Schedule A 2 mg LY2523355: 2 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day cycle.
- Schedule A 4 mg LY2524455: 4 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day cycle.
- Schedule A,C 5 mg LY2523355: Schedule A 5 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day Cycle in Part A and Part C combined.
- Schedule A 6 mg LY2523355: 6 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day cycle.
- Schedule B 8 mg LY2523355: 8 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 5, and 9 of every 21-day cycle.
- Schedule B 10 mg LY2523355: 10 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 5, and 9 of every 21-day cycle.
- Schedule B 12 mg LY2523355: 12 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1,5, and 9 of every 21-day cycle.
- Schedule B 14 mg 2523355: 14 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 5, and 9 of every 21-day cycle.
- Schedule B 16 mg LY2523355: 16 mg/m²/day was inadvertently given to a participant.
Arm/Group | Schedule A 2 mg LY2523355 | Schedule A 4 mg LY2524455 | Schedule A,C 5 mg LY2523355 | Schedule A 6 mg LY2523355 | Schedule B 8 mg LY2523355 | Schedule B 10 mg LY2523355 | Schedule B 12 mg LY2523355 | Schedule B 14 mg 2523355 | Schedule B 16 mg LY2523355
Number analyzed (Participants) | 3 | 1 | 7 | 6 | 5 | 3 | 4 | 2 | 1
nanograms per milliliter (ng/mL) | 198 (1410) | 895 (NA) — N=1, individual data presented | 240 (420) | 391 (254) | 169 (47) | 354 (66) | 254 (18) | NA (NA) — N=2,individual values presented (263 and 657), no CV calculated due to N of 2 | 17,000 (NA) — N=1, individual data presented

4. Secondary Outcome: Pharmacokinetics, Maximum Plasma Concentration (Cmax), Multiple Dose
Description: The maximum plasma concentration (Cmax) was the maximum plasma concentration obtained from the plasma concentration versus time curves of LY2523355. Multiple dose LY2523355 plasma Cmax values are shown at each dose level for both schedules of administration (Day 3 of Cycle 1 for the Day 1, 2, and 3 schedule of administration and Day 9 of Cycle 1 for the Days 1, 5, and 9 schedule of administration). The maximum plasma concentration (Cmax) was the maximum plasma concentration obtained from the plasma concentration versus time curves of LY2523355 were calculated to assess intra and intercycle variability, depending on dosage cycle.
Time Frame: Days 3 (Parts A or C) or 9 (Part B), Cycle 1: Predose, 1 hour (hr), 2 hr, 3 hr, 4 hr, 6 hr, 8, hr, 12 hr, 24 hr, 48 hr, 72 hr postdose
Population: Participants who received more than one dose of LY2523355 with evaluable pharmacokinetic data, Schedules A,B,C.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Schedule A Day 3 2 mg LY2523355: 2 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day cycle
- Schedule A Day 3 4 mg LY2523355: 4 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day cycle
- Schedule A/C Day 3 5 mg LY2523355: 5 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day cycle.
- Schedule A Day 3 6 mg LY2523355: 6 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day cycle.
- Schedule B Day 9 8 mg LY2523355: 8 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 5, and 9 of every 21-day cycle
- Schedule B Day 9 10 mg LY2523355: 10 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 5, and 9 of every 21-day cycle
- Schedule B Day 9 12 mg LY2523355: 12 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day Cycle in Part A, Part B and Part C.
- Schedule B Day 9 14 mg LY2523355: 14 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1,5, and 9 of every 21-day cycle
Arm/Group | Schedule A Day 3 2 mg LY2523355 | Schedule A Day 3 4 mg LY2523355 | Schedule A/C Day 3 5 mg LY2523355 | Schedule A Day 3 6 mg LY2523355 | Schedule B Day 9 8 mg LY2523355 | Schedule B Day 9 10 mg LY2523355 | Schedule B Day 9 12 mg LY2523355 | Schedule B Day 9 14 mg LY2523355
Number analyzed (Participants) | 3 | 1 | 9 | 5 | 3 | 3 | 2 | 1
nanograms per milliliter (ng/mL) | 43.1 (46) | 2440 (NA) — N=1, Individual parameter listed | 439 (391) | 187 (69) | 155 (139) | 283 (23) | NA (NA) — N=2. individual numbers listed: 300;14,490 | 892 (NA) — N=1,Individual parameters listed

5. Secondary Outcome: Pharmacokinetics, Area Under the Concentration Versus Time Curve (AUC), Single Dose
Description: The AUC(0-24) was calculated from area under the plasma concentration versus time curves of LY2523355 from time zero to 24 hours.
  The AUC(0-inf) was calculated from area under the plasma concentration versus time curves of LY2523355 from time zero to infinity.
  Single dose LY2523355 AUC values are shown for each dose level for Day 1 of Cycle 1 for both schedules of administration. When only individual participant parameters are available or N=2, for a given dose, the AUC CV is not calculated for that dose group and is not presented (4 milligrams per meter squared per day [mg/m^2/day], 14 mg/m^2/day, 12 mg/m^2/day and 16 mg/m^2/day). Individual data will be presented.
Time Frame: Day 1, Cycle 1: Predose, 1 hour (hr), 2 hr, 3 hr, 4 hr, 6 hr, 8, hr, 12 hr, 24 hr, 48 hr, 72 hr postdose
Population: Participants who received one dose of LY2523355 on Day 1 of Cycle 1 with evaluable pharmacokinetic data to enable calculation of the LY2523355 AUC on Day 1 of Cycle 1.Schedule A,C data was combined for 5 mg, 2 participants received and incorrect dose of 6 mg and 16 mg are included in data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanagram hours per milliliter (ng*h/mL)
Groups:
- Schedule A Day 1 2 mg LY2523355: 2 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day cycle
- Schedule A Day 1 4 mg LY2524455: 4 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day cycle
- Schedule A,C Day 1 5 mg LY2523355: 5 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day Cycle in Part A and Part C combined.
- Schedule A Day 1 6 mg LY2523355: 6 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day cycle
- Schedule B Day 1 8 mg LY2523355: 8 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 5, and 9 of every 21-day cycle.
- Schedule B Day 1 10 mg LY2523355: 10 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 5, and 9 of every 21-day cycle.
- Schedule B Day 1 12 mg LY2523355: 12 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1,5, and 9 of every 21-day cycle.
- Schedule B Day 1 14 mg 2523355: 14 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 5, and 9 of every 21-day cycle.
- Schedule B Day 1 16 mg LY2523355: 16 mg/m²/day was inadvertently given to a participant.
Arm/Group | Schedule A Day 1 2 mg LY2523355 | Schedule A Day 1 4 mg LY2524455 | Schedule A,C Day 1 5 mg LY2523355 | Schedule A Day 1 6 mg LY2523355 | Schedule B Day 1 8 mg LY2523355 | Schedule B Day 1 10 mg LY2523355 | Schedule B Day 1 12 mg LY2523355 | Schedule B Day 1 14 mg 2523355 | Schedule B Day 1 16 mg LY2523355
Number analyzed (Participants) | 3 | 1 | 9 | 5 | 3 | 3 | 2 | 2 | 1
nanagram hours per milliliter (ng*h/mL)
  The AUC(0-24) | 278 (209) | 3420 (NA) — N=1, individual data presented | 473 (163) | 613 (92) | 469 (22) | 1060 (31) | 746 (46) | NA (NA) — N=2, no CV, individual values presented: 814,1670 | 8770 (NA) — N=1, individual data presented
  The AUC(0-inf) | 229 (191) | 3490 (NA) — N=1, individual data presented | 537 (157) | 675 (86) | 608 (28) | 1530 (29) | 970 (55) | NA (NA) — N=2, no CV, individual values presented: 1150;2270 | 9200 (NA) — N=1, individual data presented

6. Secondary Outcome: Pharmacokinetics, Area Under the Concentration Versus Time (AUC), Multiple Dose
Description: The AUC(0-24) was calculated from area under the plasma concentration versus time curves of LY2523355 from time zero to 24 hours.
  The AUC(0-inf) was calculated from area under the plasma concentration versus time curves of LY2523355 from time zero to infinity..
  Multiple dose LY2523355 AUC values are shown at each dose level for both schedules of administration (Day 3 of Cycle 1 for the Day 1, 2, and 3 schedule of administration and Day 9 of Cycle 1 for the Days 1, 5, and 9 schedule of administration). When only individual participant parameters are available or N=2, for a given dose, the AUC CV is not calculated for that dose group and is not presented (4 milligrams per meter squared per day [mg/m^2/day], 12 mg/m^2/day, and 14 mg/m^2/day). Individual data will be presented.
Time Frame: Days 3 (Parts A or C) or 9 (Part B):Predose, 1 hour (hr), 2 hr, 3 hr, 4 hr, 6 hr, 8, hr, 12 hr, 24 hr 48 hr, 72 hr postdose
Population: Participants who received more than one dose of LY2523355 with evaluable pharmacokinetic data on Cycle 1 Day 3 or Day 9, schedule dependent.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms hours per milliliter (ng*h/mL)
Arm/Group | Schedule A Day 3 2 mg LY2523355 | Schedule A Day 3 4 mg LY2523355 | Schedule A/C Day 3 5 mg LY2523355 | Schedule A Day 3 6 mg LY2523355 | Schedule B Day 9 8 mg LY2523355 | Schedule B Day 9 10 mg LY2523355 | Schedule B Day 9 12 mg LY2523355 | Schedule B Day 9 14 mg LY2523355
Number analyzed (Participants) | 3 | 1 | 9 | 6 | 3 | 3 | 2 | 1
nanograms hours per milliliter (ng*h/mL)
  AUC(0-24) | 134 (38) | 2540 (NA) — Individual parameter listed | 696 (126) | 624 (66) | 623 (81) | 844 (14) | NA (NA) — N= 2, individual parameter listed: 1200;6380 | 2910 (NA) — Individual parameter listed
  AUC(0-inf), | 187 (45) | 3120 (NA) — Individual parameter listed | 992 (117) | 990 (107) | 834 (98) | 1050 (8) | NA (NA) — N= 2, individual parameter listed: 1560; 6390 | 4120 (NA) — Individual parameter listed

7. Secondary Outcome: Percentage of Participants With a Response for Acute Myelogenous Leukemia Using The Revised International Working Group Criteria
Description: Response rate for participants with acute myelogenous leukemia include the proportion of participants who achieved a morphologic complete remission, morphologic complete remission with incomplete blood count recovery, cytogenetic complete remission, molecular complete remission, or partial remission. The Revised International Working Group Criteria was used to determine response rate for participants with acute myelogenous leukemia.
Time Frame: Baseline up to disease progression or discontinuation (up to 213 days)
Population: Participants with acute myelogenous leukemia who received at least one dose of study medication (LY2523355).
Measure: Number; unit: percentage of responders
Groups:
- Schedule A LY2523355 Days 1, 2, and 3: Starting dose was 2 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day Cycle.
  Four of the 10 participants enrolled in Part A escalated from their initial dose after the first cycle (3 participants escalated from 2 to 4 mg/m^2/day and 1 participant escalated from 5 to 6 mg/m^2/day).
- Schedule B LY2523355 Days 1, 5, and 9: Starting dose was 8 mg/m^2/day administered by a 1-hour IV infusion on Days 1, 5, and 9 of every 21-day Cycle.
  Five of the 15 participants enrolled in Part B escalated from their initial dose after the first cycle (2 participants escalated from 8 to 10 mg/m^2/day, 1 participant escalated from 8 to 12 mg/m^2/day, 1 participant escalated from 10 to 12 mg/m^2/day, and 1 participant escalated from 12 to 14 mg/m^2/day).
- Schedule C LY2523355 Days 1, 2, and 3: Starting dose was 5 mg/m^2/day administered by a 1-hour IV infusion on Days 1, 5, and 9 of every 21-day Cycle.
  No participants in Part C escalated from their initial dose.
Arm/Group | Schedule A LY2523355 Days 1, 2, and 3 | Schedule B LY2523355 Days 1, 5, and 9 | Schedule C LY2523355 Days 1, 2, and 3
Number analyzed (Participants) | 5 | 9 | 8
percentage of responders | 0.0 | 11.1 | 12.5

8. Secondary Outcome: Response Rates for Chronic Myelogenous Leukemia in Blast Crisis (Complete Hematologic Response, no Evidence of Leukemia, Return to Chronic Phase)
Description: Response rate for participants with chronic myelogenous leukemia in blast crisis include the proportion of participants who achieved a complete hematologic response, had no evidence of leukemia, or had returned to chronic phase. The criteria outlined in Cohen 2005 (Cohen MH, Johnson JR, Pazdur R. 2005. U.S. Food and Drug Administration Drug Approval Summary: conversion of imatinib mesylate (STI571; Gleevec) tablets from accelerated approval to full approval. Clin Cancer Res. 11(1):12-19.) was used to determine response rate for participants with chronic myelogenous leukemia in blast crisis.
Time Frame: Baseline up to disease progression or discontinuation (up to 213 days)
Population: Participants with chronic myelogenous leukemia in blast crisis who received at least one dose of study medication (LY2523355).
Measure: Number; unit: percentage of responders
Groups:
- Schedule A LY2523355 Days 1, 2, and 3: Starting dose was 2 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 5, and 9 of every 21-day Cycle.
  Four of the 10 participants enrolled in Part A escalated from their initial dose after the first cycle (3 participants escalated from 2 to 4 mg/m^2/day and 1 participant escalated from 5 to 6 mg/m^2/day).
Arm/Group | Schedule A LY2523355 Days 1, 2, and 3 | Schedule B LY2523355 Days 1, 5, and 9 | Schedule C LY2523355 Days 1, 2, and 3
Number analyzed (Participants) | 0 | 1 | 0
percentage of responders |  | 0 |

9. Secondary Outcome: Response Rate (Percentage) for Acute Lymphoblastic Leukemia Using The Revised International Working Group Criteria
Description: Response rate for participants with acute lymphoblastic leukemia include the proportion of participants who achieved a morphologic complete remission, morphologic complete remission with incomplete blood count recovery, cytogenetic complete remission, molecular complete remission, or partial remission. The Revised International Working Group Criteria was used to determine response rate for participants with acute lymphoblastic leukemia by early treatment assessment, morphologic leukemia-free state (less than 5% blasts in an aspirate sample with marrow spicules and with a count of at least 200 nucleated cells) and morphologic complete remission (and have an absolute neutrophil count of more than 1000 per microliter and platelets of 100,000 per microliter.
Time Frame: Baseline up to disease progression or discontinuation (up to 213 days)
Population: Participants with acute lymphoblastic leukemia who received at least one dose of study medication (LY2523355).
Measure: Number; unit: percentage of responders
Arm/Group | Schedule A LY2523355 Days 1, 2, and 3 | Schedule B LY2523355 Days 1, 5, and 9 | Schedule C LY2523355 Days 1, 2, and 3
Number analyzed (Participants) | 4 | 0 | 0
percentage of responders | 25.0 |  |

10. Other Pre Specified Outcome: Death of Participants on Study up to the Follow-up Period
Description: The number of participants who died through the follow-up period of the study. This does not include the outcomes for the two participants who died while on treatment through Cycle 2 as captured in the Participant Flow Table.
  A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline up to end of treatment follow-up (up to 213 days)
Population: Participants who received at least one dose of study medication (LY2523355).
Measure: Count of Participants; unit: Participants
Groups:
- Schedule LY2523355 Days 1, 2, and 3: Starting dose was 2 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 5, and 9 of every 21-day Cycle.
  Four of the 10 participants enrolled in Part A escalated from their initial dose after the first cycle (3 participants escalated from 2 to 4 mg/m^2/day and 1 participant escalated from 5 to 6 mg/m^2/day).
Arm/Group | Schedule LY2523355 Days 1, 2, and 3 | Schedule B LY2523355 Days 1, 5, and 9 | Schedule C LY2523355 Days 1, 2, and 3
Number analyzed (Participants) | 10 | 15 | 8
Participants | 1 | 4 | 0

ADVERSE EVENTS:
Description: AEs were listed and the incidence summarized by study part, assigned dose level. For participants that were escalated within their dose group, AEs were counted for both dose levels. Participants who escalated dose are represented in 2 columns.
Groups:
- Cohort 1 LY2523355 2 mg/m^2/Day, Days 1, 2, and 3: Dose was 2 milligrams per meter squared per day (mg/m^2/day) administered by a 1-hour intravenous (IV) infusion on Days 1, 2, and 3 of every 21-day Cycle.
- Cohort 1 LY2523355 4 mg/m^2/Day, Days 1, 2, and 3: Dose was 4 mg/m^2/day administered by a 1-hour IV infusion on Days 1, 2, and 3 of every 21-day Cycle.
- Cohort 1 LY2523355 5 mg/m^2/Day, Days 1, 2, and 3; Cohort 3 LY2523355 5 mg/m^2/Day, Days 1, 2, and 3: Dose was 5 mg/m^2/day administered by a 1-hour IV infusion on Days 1, 2, and 3 of every 21-day Cycle.
- Cohort 1 LY2523355 6 mg/m^2/Day, Days 1, 2, and 3: Dose was 6 mg/m^2/day administered by a 1-hour IV infusion on Days 1, 2, and 3 of every 21-day Cycle.
- Cohort 2 LY2523355 8 mg/m^2/Day, Days 1, 5, and 9: Dose was 8 mg/m^2/day administered by a 1-hour IV infusion on Days 1, 5, and 9 of every 21-day Cycle.
- Cohort 2 LY2523355 10 mg/m^2/Day, Days 1, 5, and 9: Dose was 10 mg/m^2/day administered by a 1-hour IV infusion on Days 1, 5, and 9 of every 21-day Cycle.
- Cohort 2 LY2523355 12 mg/m^2/Day, Days 1, 5, and 9: Dose was 12 mg/m^2/day administered by a 1-hour IV infusion on Days 1, 5, and 9 of every 21-day Cycle.
- Cohort 2 LY2523355 14 mg/m^2/Day, Days 1, 5, and 9: Dose was 14 mg/m^2/day administered by a 1-hour IV infusion on Days 1, 5, and 9 of every 21-day Cycle.
Arm/Group | Cohort 1 LY2523355 2 mg/m^2/Day, Days 1, 2, and 3 | Cohort 1 LY2523355 4 mg/m^2/Day, Days 1, 2, and 3 | Cohort 1 LY2523355 5 mg/m^2/Day, Days 1, 2, and 3 | Cohort 1 LY2523355 6 mg/m^2/Day, Days 1, 2, and 3 | Cohort 2 LY2523355 8 mg/m^2/Day, Days 1, 5, and 9 | Cohort 2 LY2523355 10 mg/m^2/Day, Days 1, 5, and 9 | Cohort 2 LY2523355 12 mg/m^2/Day, Days 1, 5, and 9 | Cohort 2 LY2523355 14 mg/m^2/Day, Days 1, 5, and 9 | Cohort 3 LY2523355 5 mg/m^2/Day, Days 1, 2, and 3
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/4 | 1/2 | 3/5 | 2/4 | 1/5 | 3/7 | 3/4 | 4/8
Other Adverse Events (participants affected / at risk) | 3/3 | 3/4 | 2/2 | 5/5 | 3/4 | 5/5 | 7/7 | 4/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 LY2523355 2 mg/m^2/Day, Days 1, 2, and 3 (N=3) | Cohort 1 LY2523355 4 mg/m^2/Day, Days 1, 2, and 3 (N=4) | Cohort 1 LY2523355 5 mg/m^2/Day, Days 1, 2, and 3 (N=2) | Cohort 1 LY2523355 6 mg/m^2/Day, Days 1, 2, and 3 (N=5) | Cohort 2 LY2523355 8 mg/m^2/Day, Days 1, 5, and 9 (N=4) | Cohort 2 LY2523355 10 mg/m^2/Day, Days 1, 5, and 9 (N=5) | Cohort 2 LY2523355 12 mg/m^2/Day, Days 1, 5, and 9 (N=7) | Cohort 2 LY2523355 14 mg/m^2/Day, Days 1, 5, and 9 (N=4) | Cohort 3 LY2523355 5 mg/m^2/Day, Days 1, 2, and 3 (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (5)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 LY2523355 2 mg/m^2/Day, Days 1, 2, and 3 (N=3) | Cohort 1 LY2523355 4 mg/m^2/Day, Days 1, 2, and 3 (N=4) | Cohort 1 LY2523355 5 mg/m^2/Day, Days 1, 2, and 3 (N=2) | Cohort 1 LY2523355 6 mg/m^2/Day, Days 1, 2, and 3 (N=5) | Cohort 2 LY2523355 8 mg/m^2/Day, Days 1, 5, and 9 (N=4) | Cohort 2 LY2523355 10 mg/m^2/Day, Days 1, 5, and 9 (N=5) | Cohort 2 LY2523355 12 mg/m^2/Day, Days 1, 5, and 9 (N=7) | Cohort 2 LY2523355 14 mg/m^2/Day, Days 1, 5, and 9 (N=4) | Cohort 3 LY2523355 5 mg/m^2/Day, Days 1, 2, and 3 (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (4)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (7)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
Before MTD could be determined for Part B (Days 1, 5, and 9 of a 21-day cycle), this study was paused for futility analysis. The decision was made to close the study because of evident toxicity and lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days